CLINICAL TRIAL: NCT02167516
Title: Efficacy and Safety of Xinfeng Capsule in the Treatment of Knee Osteoarthritis (KOA) :A Randomized, Double-blind, Double-dummy, Multi-center Trial
Brief Title: A Clinical Study of Xin'an Medicine in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Liu Jian, professor，Chief Physician, The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1301042211
Record Dates: First submitted 2014-06-15; First posted 2014-06-19 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Knee Osteoarthritis
Keywords: Xinfeng capsule; Knee osteoarthritis; Randomized controlled trials; Double-blind
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine; xinfeng

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xinfeng capsule (Experimental): Xinfeng capsule:Three each time, 3 times a day, Oral,for 4 weeks placebo(for glucosamine sulfate capsule): One each time, 3 times a day, Oral,for 4 weeks
  Interventions: Drug: Xinfeng capsule
- glucosamine sulfate capsule (Active Comparator): glucosamine sulfate capsule: One each time, 3 times a day, Oral,for 4 weeks placebo(for Xinfeng capsule): Three each time, 3 times a day, Oral,for 4 weeks
  Interventions: Drug: glucosamine sulfate

INTERVENTIONS:
Drug: glucosamine sulfate — glucosamine sulfate capsule: One each time, 3 times a day, Oral,for 4 weeks placebo(for Xinfeng capsule): Three each time, 3 times a day, Oral,for 4 weeks
  Arms: glucosamine sulfate capsule
Drug: Xinfeng capsule — Xinfeng capsule:Three each time, 3 times a day, Oral,for 4 weeks placebo(for glucosamine sulfate capsule): One each time, 3 times a day, Oral,for 4 weeks
  Arms: Xinfeng capsule

SUMMARY:
Complementary and alternative medicine has been employed over thousands of years to relieve knee Osteoarthritis (OA) pain. Xinfeng Capsule, a patent Chinese herbal medicine, has been used in the treatment of Knee Osteoarthritis (KOA) Some studies involving animal subjects may explored its mechanism. However, presently, there is a lack of large-sample, multicenter, randomized, controlled trials to evaluate the effects of Xinfeng Capsule treated for KOA. Therefore, the investigators designed a randomized, placebo-controlled, double-blind, multicenter trial to evaluate the effectiveness and safety of Xinfeng Capsule in the treatment of KOA.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the American College of Rheumatology (ACR) 1995 revised criteria for KOA.
* Participants must be aged between 40 and 75 years.
* Participants shall not take non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroids during the 7 days prior to screening.
* Participants shall not take Chinese medicine for the treatment of KOA during the 7 days prior to screening.
* Joint function in the I-III, X-ray stage in the I-III.
* All participants shall agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Patients whose joint clearance is significantly narrow or joint bone bridge connection is formed between a bony rigidity.
* Patients who have knee cancer, rheumatoid arthritis, tuberculosis, acute purulent or intra-articular fractures.
* Persons have obvious inside and outside of the knee varus deformity and a history of limb vascular nerve injury .
* Patients with severe cardiovascular, brain, lung, liver, kidney, or hematopoietic diseases.
* Pregnant women or breastfeeding mothers or individuals with known psychiatric disorders.
* Patients who are hypersensitive to the trial medication.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index (WOMAC) | up to week 4

SECONDARY OUTCOMES:
Arthritis pain assessment using the Visual Analog scale (VAS) | baseline,week2,week4
KOA severity using the Lequesne MG score | baseline,week2,week4
Erythrocyte sedimentation rate (ESR), C-reactive protein, alkaline phosphatase (ALP), superoxide dismutase (SOD) and serum calcium | baseline,week4
Bilateral femoral bone mineral density. | baseline,week4
Health assessment of the patient refer to the MOS item short from health survey (SF-36) | baseline,week4

CONTACTS AND LOCATIONS:
Overall Officials: Jian Liu, Principal Investigator — The First Affiliated Hospital of Anhui University of Chinese Medicine
Locations (3):
- China (3):
  - the First Affiliated Hospital of Anhui University of Chinese Medicine, Hefei, Anhui
  - The Taihe County Hospital of Chinese Medicine, Taihe Chengguanzhen, Anhui
  - The Tianchang City Hospital of Chinese Medicine, Tianchang, Anhui